CLINICAL TRIAL: NCT02517866
Title: A Prospective Study of Azilsartan Medoxomil in the Treatment of Patients With Essential Hypertension and Type 2 Diabetes in Asia
Brief Title: Azilsartan Medoxomil in the Treatment of Essential Hypertension and Type 2 Diabetes in Asia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZI-P4-002; U1111-1156-8501 (Registry Identifier: WHO)
Record Dates: First submitted 2015-06-24; First posted 2015-08-07 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2018-10

CONDITIONS: Essential Hypertension; Type 2 Diabetes Mellitus
Keywords: Drug therapy
MeSH Terms: conditions — Essential Hypertension; Diabetes Mellitus, Type 2 | interventions — azilsartan medoxomil; azilsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azilsartan medoxomil (Experimental): Azilsartan medoxomil 40 mg, tablets, orally, once, daily, for 12 weeks. Azilsartan medoxomil dose may be increased to 80 mg once daily if blood pressure has not reach BP goal of <140/85 mmHg at Week 6.
  Interventions: Drug: Azilsartan Medoxomil

INTERVENTIONS:
Drug: Azilsartan Medoxomil — Azilsartan medoxomil tablets
  Other Names: Edarbi®

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of azilsartan medoxomil (AZM) in Asian adult participants with both essential hypertension and type 2 diabetes.

DETAILED DESCRIPTION:
The drug being tested in this study is called azilsartan medoxomil. Azilsartan medoxomil is being tested to treat people who have essential hypertension and type 2 diabetes mellitus (T2DM). This study will look at the blood pressure of people who take azilsartan medoxomil in addition to standard care for T2DM.

The study will enroll approximately 380 patients. All participants will receive azilsartan medoxomil 40 mg tablets to be administered orally, once a day, for 12 weeks. If a participant's blood pressure (BP) has not reached BP goal of <140/85 mmHg at week 6, azilsartan medoxomil dose will be up-titrated to 80 mg daily.

All participants will be asked to take one tablet at the same time each day throughout the study.

This multi-center trial will be conducted in Asia. The overall time to participate in this study is 14 weeks. Participants will make multiple visits to the clinic, and will be contacted by 14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has type 2 diabetes mellitus (T2DM) with essential hypertension.
4. T2DM participants are either treated by stable life style intervention or by oral antidiabetic drugs (OADs) that are stable, including no dose adjustment within 12 weeks before baseline.
5. Is male or female and aged 18 to 75 years, inclusive.
6. Uncontrolled hypertension (systolic blood pressure ≥140 mmHg to <180 mmHg, or diastolic blood pressure ≥85 mmHg and <110 mmHg at screening and baseline.
7. Has screening glycosylated hemoglobin (HbA1C) <9.5%.
8. Female participants must be either of non-childbearing potential, ie, surgically sterilized (defined as having undergone hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy; tubal ligation alone is not considered sufficient) or one year after the last menstrual period; or, if of childbearing potential and participant is sexually active with a nonsterilized male partner, must agree to use routinely adequate contraception from signing of informed consent throughout the duration of study.

Exclusion Criteria:

1. Has systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg despite concurrent treatment with three antihypertensive medications from different classes at adequate doses including a diuretic.
2. Has type 1 or poorly controlled type 2 diabetes mellitus, defined as HbA1c ≥9.5% at screening.
3. Is treated with OADs has not been on stable treatment including no dose change of their OADs for at least 12 weeks prior to baseline.
4. Has been previously treated with azilsartan medoxomil (AZM) or azilsartan.
5. Has secondary hypertension of any etiology (eg, renovascular disease, pheochromocytoma, Cushing's syndrome).
6. Has congestive heart failure (New York Heart Association class III or IV), clinically relevant cardiac arrhythmias (as determined by the investigator's clinical judgment on a participant-by-participant basis), severe obstructive coronary artery disease.
7. Has participated in a clinical trial including interventional and observational studies, or received any investigational compound currently or 30 days prior to screening.
8. Has severe renal impairment (based on estimated glomerular filtration rate [GFR] <30 mL/min/1.73m^2) at Screening.
9. Has hyperkalemia defined as serum potassium >5.0 mEq/L.
10. Has an alanine aminotransferase (ALT) level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice at screening.
11. Has any clinically relevant disease (eg malignancy, neurological, hepatic abnormalities) and/or significant abnormal laboratory findings (past or present), which, in the opinion of the investigator, may put the participant at risk because of participation in the study.
12. Is taking prohibited medications including lithium and aliskiren (refer to Edarbi® product insert).
13. Has known hypersensitivity to any excipients or angiotensin converting enzyme inhibitor (ACEIs)/ angiotensin receptor blockers (ARBs).
14. Has prior angioedema due to an ACE inhibitor or ARB.
15. Breast feeding or pregnant women or women who are intending to become pregnant before, during or within 1 month after participating in the study; or intending to donate ova during such time period, or refusal to submit to a urine test to rule out pregnancy prior to enrolment and at end of study.
16. Have a history of alcohol abuse, drug abuse or illegal drug addiction within the 6 months prior to signing the informed consent.
17. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (11):
- Hong Kong, Hong Kong, China
- Taiwan (6):
  - Changhua County
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan
- Thailand (4):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
  - Pathum Thani

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 34 investigative sites in Hong Kong, Taiwan and Thailand from 13 July 2015 to 25 November 2016.
Pre-assignment Details: Participants with a diagnosis of essential hypertension and type 2 diabetes mellitus (T2DM) were enrolled to receive azilsartan medoxomil at a starting dose of 40 mg increased to 80 mg if blood pressure of <140/85 mmHg was not achieved at Week 6.
Groups:
- Azilsartan Medoxomil (Switched): Azilsartan medoxomil 40 mg, tablets, orally, once, daily, for 12 weeks. Azilsartan medoxomil dose may be increased to 80 mg once daily if blood pressure has not reach BP goal of <140/85 mmHg at Week 6. Switched includes participants who switched from their baseline hypertension therapy to azilsartan medoxomil.
- Azilsartan Medoxomil (Add-On): Azilsartan medoxomil 40 mg, tablets, orally, once, daily, for 12 weeks. Azilsartan medoxomil dose may be increased to 80 mg once daily if blood pressure has not reach BP goal of <140/85 mmHg at Week 6. Add-On includes participants who added azilsartan medoxomil to their baseline hypertension therapy.
- Azilsartan Medoxomil (Treatment-Naïve): Azilsartan medoxomil 40 mg, tablets, orally, once, daily, for 12 weeks. Azilsartan medoxomil dose may be increased to 80 mg once daily if blood pressure has not reach BP goal of <140/85 mmHg at Week 6. Treatment-naïve includes participants never treated with antihypertensive therapy or participants who did not receive hypertension therapy for at least 4 weeks prior to screening.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil (Switched) | Azilsartan Medoxomil (Add-On) | Azilsartan Medoxomil (Treatment-Naïve)
Started | 289 | 90 | 1
Completed | 269 | 84 | 1
Not Completed | 20 | 6 | 0
Not completed — Pretreatment Event/Adverse Event | 9 | 2 | 0
Not completed — Significant Protocol Deviation | 4 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Voluntary Withdrawal | 2 | 2 | 0
Not completed — Investigator Decision | 2 | 1 | 0
Not completed — Reason not specified | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who took at least 1 dose of azilsartan medoxomil.
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 380
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.77)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years old | 221
  >=65 to <75 years old | 159
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197
  Male | 183
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 380
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan, Province Of China | 139
  Thailand | 219
  Hong Kong | 22
Height [Mean (Standard Deviation); unit: cm] | 161.1 (9.57)
Weight [Mean (Standard Deviation); unit: kg] — Population: Here number analyzed is the number of participants who were evaluated for weight at baseline.
  kg
    number analyzed (Participants) | 374
    (all) | 72.04 (15.072)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Here number analyzed is the number of participants who were evaluated for BMI at baseline.
  kg/m^2
    number analyzed (Participants) | 374
    (all) | 27.64 (4.354)
Smoking history [Count of Participants; unit: Participants]
  The participant has never smoked | 279
  The participant is an ex-smoker | 75
  The participant is a current smoker | 26
Baseline Antihypertensive Treatment Status [Number; unit: participants] — Participants were counted more than once according to the antihypertensive treatment status. Antihypertensive treatment includes Angiotensin Converting Enzyme (ACE) inhibitor, Angiotensin Receptor Blocker (ARB), Calcium Channel Blocker (CCB), Thiazides and/or other treatments.
  participants
    Treated with ACE inhibitor or ARB before Baseline | 202
    Treated with CCB before Baseline | 112
    Treated with Thiazide before Baseline | 30
    Other | 121
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: mmoL/moL] — Population: Only 374 participants were evaluated for this baseline characteristic.
  mmoL/moL
    number analyzed (Participants) | 374
    (all) | 7.00 (0.875)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Blood Pressure (BP) <140/85 mmHg (Systolic BP <140 mmHg and Diastolic BP <85 mmHg) by Clinic-Measured Sitting BP at Week 12
Description: Three serial BP measurements were determined while the participant was seated, with a sphygmomanometer.
Time Frame: Week 12
Population: Full analysis set (FAS) included all participants who took at least 1 dose of azilsartan medoxomil. Missing data was computed using last observation carried forward (LOCF) method. Here, number of participants analyzed is the total number of participants who were evaluable for this outcome measure.
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil (Switched) | Azilsartan Medoxomil (Add-On)
Number analyzed (Participants) | 276 | 85
percentage of participants | 59.8 [43.40 to 63.08] | 65.9 [44.07 to 75.70]

2. Secondary Outcome: Percentage of "Treatment-Naïve" Participants Reaching BP <140/85 mmHg
Description: Treatment-naïve participants are defined as participants who have not received anti-hypertensive treatment for at least four weeks prior to screening. At each visit 3 serial BP measurements were determined while the participant was seated, with a sphygmomanometer.
Time Frame: Up to Week 12
Population: FAS included all participants who took at least 1 dose of azilsartan medoxomil.
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil (Treatment-Naïve)
Number analyzed (Participants) | 1
percentage of participants | 0.0 [NA to NA] — CI was not calculated as there was only one participant in this group.

3. Secondary Outcome: Percentage of Participants Treated With Calcium Channel Blocker (CCB) Before Baseline Reaching BP<140/85 mmHg
Description: At each visit three serial BP measurements were determined while the participant was seated, with a sphygmomanometer.
Time Frame: Weeks 6 and 12
Population: FAS included all participants who took at least 1 dose of azilsartan medoxomil. Missing data was computed using LOCF method. Here, number of participants analyzed is the participants who received CCB before baseline and are evaluable for this outcome measure.
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 109
percentage of participants
  Week 6 | 57.8 [45.36 to 71.12]
  Week 12 | 52.3 [39.75 to 65.08]

4. Secondary Outcome: Percentage of Participants Treated With Angiotensin Converting Enzyme (ACE) Inhibitors or Other Angiotensin Receptor Blockers (ARBs) Before Baseline Reaching BP <140/85 mmHg
Description: At each visit 3 serial BP measurements were determined while the participant was seated, with a sphygmomanometer.
Time Frame: Weeks 6 and 12
Population: FAS included all participants who took at least 1 dose of azilsartan medoxomil. Missing data was computed using LOCF method. Here, number of participants analyzed is the participants who received ACE inhibitors or other ARBs before baseline and are evaluable for this outcome measure.
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 193
percentage of participants
  Week 6 | 63.7 [44.83 to 68.92]
  Week 12 | 63.7 [44.73 to 69.01]

5. Secondary Outcome: Percentage of Participants Treated With Thiazides Before Baseline Reaching BP <140/85 mmHg
Description: At each visit three serial BP measurements were determined while the participant was seated, with a sphygmomanometer.
Time Frame: Weeks 6 and 12
Population: FAS included all participants who took at least 1 dose of azilsartan medoxomil. Missing data was computed using LOCF method. Here, number of participants analyzed is the participants who received thiazides before baseline and are evaluable for this outcome measure.
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 29
percentage of participants
  Week 6 | 79.3 [45.97 to 89.46]
  Week 12 | 86.2 [43.81 to 97.18]

6. Secondary Outcome: Percentage of "Treatment-Naïve" Participants Reaching BP <130/80 mmHg
Description: as for outcome 2
Time Frame: Up to Week 12
Population: FAS included all participants who took at least 1 dose of azilsartan medoxomil.
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil (Treatment-Naïve)
Number analyzed (Participants) | 1
percentage of participants | 0.0 [NA to NA] — CI was not calculated as there was only one participant in this group.

7. Secondary Outcome: Percentage of Participants Treated With CCB Before Baseline Reaching BP <130/80 mmHg
Description: At each visit 3 serial BP measurements were determined while the participant was seated, with a sphygmomanometer.
Time Frame: Weeks 6 and 12
Population: as for outcome 3
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 109
percentage of participants
  Week 6 | 26.6 [14.73 to 36.50]
  Week 12 | 27.5 [15.73 to 37.10]

8. Secondary Outcome: Percentage of Participants Treated With ACE Inhibitors or Other ARBs Before Baseline Reaching BP <130/80 mmHg
Description: At each visit 3 serial BP measurements were determined while the participant was seated, with a sphygmomanometer.
Time Frame: Weeks 6 and 12
Population: as for outcome 4
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 193
percentage of participants
  Week 6 | 31.1 [10.05 to 33.20]
  Week 12 | 35.2 [12.18 to 37.37]

9. Secondary Outcome: Percentage of Participants Treated With Thiazides Before Baseline Reaching BP <130/80 mmHg
Description: At each visit 3 serial BP measurements were determined while the participant was seated, with a sphygmomanometer.
Time Frame: Weeks 6 and 12
Population: as for outcome 5
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 29
percentage of participants
  Week 6 | 41.4 [21.13 to 65.05]
  Week 12 | 51.7 [29.12 to 73.67]

10. Secondary Outcome: Percentage of Participants With Systolic Blood Pressure (SBP) <140 mmHg at Week 12
Description: Three serial BP measurements were determined while the participant was seated, with a sphygmomanometer.
Time Frame: Week 12
Population: FAS included all participants who took at least 1 dose of azilsartan medoxomil. Missing data was computed using LOCF method. Here, number of participants analyzed is the total number of participants who were evaluable for this outcome measure.
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil (Switched) | Azilsartan Medoxomil (Add-On) | Azilsartan Medoxomil (Treatment-Naïve)
Number analyzed (Participants) | 276 | 85 | 1
percentage of participants | 68.8 [57.57 to 75.78] | 70.6 [52.49 to 83.94] | 0.0 [NA to NA] — CI was not calculated as there was only one participant in this group.

11. Secondary Outcome: Percentage of Participants With Diastolic Blood Pressure (DBP) <85 mmHg at Week 12
Description: Three serial BP measurements were determined while the participant was seated, with a sphygmomanometer.
Time Frame: Week 12
Population: as for outcome 10
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil (Switched) | Azilsartan Medoxomil (Add-On) | Azilsartan Medoxomil (Treatment-Naïve)
Number analyzed (Participants) | 276 | 85 | 1
percentage of participants | 74.6 [64.86 to 81.66] | 81.2 [67.40 to 91.05] | 0.0 [NA to NA] — CI was not calculated as there was only one participant in this group.

12. Secondary Outcome: Percentage of Participants With DBP <90 mmHg at Week 12
Description: Three serial BP measurements were determined while the participant was seated, with a sphygmomanometer.
Time Frame: Week 12
Population: as for outcome 10
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil (Switched) | Azilsartan Medoxomil (Add-On) | Azilsartan Medoxomil (Treatment-Naïve)
Number analyzed (Participants) | 276 | 85 | 1
percentage of participants | 87.3 [85.11 to 95.34] | 87.1 [79.97 to 96.46] | 0.0 [NA to NA] — CI was not calculated as there was only one participant in this group.

13. Secondary Outcome: Percentage of Participants With BP <130/80 mmHg at Week 12
Description: Three serial BP measurements were determined while the participant was seated, with a sphygmomanometer.
Time Frame: Week 12
Population: as for outcome 10
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil (Switched) | Azilsartan Medoxomil (Add-On) | Azilsartan Medoxomil (Treatment-Naïve)
Number analyzed (Participants) | 276 | 85 | 1
percentage of participants | 33.7 [17.01 to 37.26] | 40.0 [18.66 to 48.66] | 0.0 [NA to NA] — CI was not calculated as there was only one participant in this group.

14. Secondary Outcome: Percentage of Participants With SBP <130 mmHg at Week 12
Description: Three serial BP measurements were determined while the participant was seated, with a sphygmomanometer.
Time Frame: Week 12
Population: as for outcome 10
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil (Switched) | Azilsartan Medoxomil (Add-On) | Azilsartan Medoxomil (Treatment-Naïve)
Number analyzed (Participants) | 276 | 85 | 1
percentage of participants | 41.3 [22.25 to 43.20] | 43.5 [20.17 to 50.31] | 0.0 [NA to NA] — CI was not calculated as there was only one participant in this group.

15. Secondary Outcome: Percentage of Participants With DBP <80 mmHg at Week 12
Description: Three serial BP measurements were determined while the participant was seated, with a sphygmomanometer.
Time Frame: Week 12
Population: as for outcome 10
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil (Switched) | Azilsartan Medoxomil (Add-On) | Azilsartan Medoxomil (Treatment-Naïve)
Number analyzed (Participants) | 276 | 85 | 1
percentage of participants | 57.6 [36.82 to 59.95] | 65.9 [41.33 to 75.07] | 0.0 [NA to NA] — CI was not calculated as there was only one participant in this group.

16. Secondary Outcome: Percentage of Participants With BP <140/90 mmHg at Week 12
Description: Three serial BP measurements were determined while the participant was seated, with a sphygmomanometer.
Time Frame: Week 12
Population: as for outcome 10
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil (Switched) | Azilsartan Medoxomil (Add-On) | Azilsartan Medoxomil (Treatment-Naïve)
Number analyzed (Participants) | 276 | 85 | 1
percentage of participants | 65.9 [52.51 to 71.04] | 68.2 [48.42 to 79.92] | 0.0 [NA to NA] — CI was not calculated as there was only one participant in this group.

17. Secondary Outcome: Change From Baseline in Trough Sitting SBP at Week 12
Description: At each visit 3 serial BP measurements were determined while the participant was seated, with a sphygmomanometer. Change from Baseline was estimated using an ANCOVA model with fixed effects, country, baseline hypertension therapy (BHT) and baseline SBP (or DBP) included as a covariate. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil (Switched) | Azilsartan Medoxomil (Add-On)
Number analyzed (Participants) | 276 | 90
mmHg | -14.1 (1.39) | -13.3 (2.12)

18. Secondary Outcome: Change From Baseline in Trough Sitting SBP at Week 12 in "Treatment-Naïve" Participants
Description: as for outcome 17
Time Frame: Baseline and Week 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan Medoxomil (Treatment-Naïve)
Number analyzed (Participants) | 1
mmHg | -7 (NA) — Standard deviation was not calculated as there was only one participant who was evaluated.

19. Secondary Outcome: Change From Baseline in DBP at Week 12
Description: At each visit 3 serial BP measurements were determined while the participant was seated, with a sphygmomanometer. Change from Baseline was estimated using an ANCOVA model with fixed effects, country, BHT and baseline SBP (or DBP) included as a covariate. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: FAS included all participants who took at least 1 dose of azilsartan medoxomil. Missing data was computed using LOCF method. Here, number of participants analyzed is the total number of participants who were analysed for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil (Switched) | Azilsartan Medoxomil (Add-On)
Number analyzed (Participants) | 276 | 85
mmHg | -4.9 (0.76) | -5.7 (1.16)

20. Secondary Outcome: Change From Baseline in DBP at Week 12 in "Treatment-Naïve" Participants
Description: as for outcome 19
Time Frame: Baseline and Week 12
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan Medoxomil (Treatment-Naïve)
Number analyzed (Participants) | 1
mmHg | 20 (NA) — Standard deviation was not calculated as there was only one participant who was evaluated.

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 14 days after the date of the last dose of study drug (up to 14 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Adverse Events are reported as per dose received.
Groups:
- Before Week 6 Azilsartan Medoxomil 40 mg: Azilsartan medoxomil 40 mg, tablets, orally, once, daily, for 6 weeks.
- After Week 6 Azilsartan Medoxomil 40 mg: Azilsartan medoxomil 40 mg, tablets, orally, once, daily, for Week 6 up to Week 12.
- After Week 6 Azilsartan Medoxomil 80 mg: Azilsartan medoxomil 80 mg, tablets, orally, once, daily, for Week 6 up to Week 12.
Arm/Group | Before Week 6 Azilsartan Medoxomil 40 mg | After Week 6 Azilsartan Medoxomil 40 mg | After Week 6 Azilsartan Medoxomil 80 mg
Serious Adverse Events (participants affected / at risk) | 4/380 | 3/258 | 1/97
Other Adverse Events (participants affected / at risk) | 0/380 | 0/258 | 0/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Before Week 6 Azilsartan Medoxomil 40 mg (N=380) | After Week 6 Azilsartan Medoxomil 40 mg (N=258) | After Week 6 Azilsartan Medoxomil 80 mg (N=97)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.